CLINICAL TRIAL: NCT01879423
Title: A Single-Dose, Open-Label, Randomized, Two-Period Crossover Study to Demonstrate the Bioequivalence of Lamotrigine Dispersible/Chewable Tablets (5mg×5) and Lamotrigine Compressed Tablet (25mg) in Healthy Chinese Male Subjects.
Brief Title: The Bioequivalence Study of Lamotrigine Dispersible/Chewable Tablets 5mg×5 Compared With Lamotrigine Compressed Tablet 25mg in Chinese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115207
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine (Lamictal) D/C 5mg*5, Crossover (Experimental): Single dose of lamotrigine dispersible/chewable (D/C)5mg*5 tablets at Day1 and Single dose of Lamotrigine Compressed 25mg*1 tablet at Day15
  Interventions: Drug: Lamotrigine Dispersible/Chewable tablets 5mg*5; Drug: Lamotrigine Compressed tablet 25mg
- Lamotrigine (Lamictal) Compressed 25mg, Crossover (Experimental): Single dose of lamotrigine compressed 25mg*1 tablet at Day1 and Single dose of lamotrigine dispersible/chewable 5mg*5 tablets at Day15
  Interventions: Drug: Lamotrigine Dispersible/Chewable tablets 5mg*5; Drug: Lamotrigine Compressed tablet 25mg

INTERVENTIONS:
Drug: Lamotrigine Dispersible/Chewable tablets 5mg*5 — Single dose of lamotrigine dispersible/chewable 5mg*5 tablets at Day1 and Single dose of Lamotrigine Compressed 25mg*1 tablet at Day15
  Other Names: Lamictal
Drug: Lamotrigine Compressed tablet 25mg — Single dose of lamotrigine compressed 25mg*1 tablet at Day1 and Single dose of lamotrigine dispersible/chewable 5mg*5 tablets at Day15
  Other Names: Lamictal

SUMMARY:
This is a single dose, open-label, randomized, two-period crossover study to demonstrate the bioequivalence of lamotrigine dispersible/chewable tablets (5mg×5) and lamotrigine compressed tablets (25mg) in healthy Chinese male subjects in fasting conditions. The safety, tolerability and pharmacokinetic profile of lamotrigine dispersible/chewable tablets will also be assessed.

DETAILED DESCRIPTION:
This is a single dose, open-label, randomized, two-period crossover study to demonstrate the bioequivalence of lamotrigine dispersible/chewable tablets (5mg×5) and lamotrigine compressed tablets (25mg) in healthy Chinese male subjects in fasting conditions. 24 healthy Chinese male subjects will be enrolled to provide data from at least 22 evaluable subjects . In Period 1, subjects will be randomized in equal numbers to be dosed with either lamotrigine dispersible/chewable 5mg×5 tablets or lamotrigine compressed tablet 25mg×1. Following a washout of at least 14 days, subjects will be crossed over in Period 2 to receive the treatment that they did not receive in Period 1.

Pharmacokinetic blood samples will be collected over 168 hours post dose. Venous blood (2 ml each) is taken immediately before dosing (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post dose to determine the lamotrigine concentration in serum. Drug concentration in serum at different time points will be determined for each subject with a validated bioanalytical method using LC/MS/MS method. The main pharmacokinetic parameters such as Cmax, tmax, AUC(0-inf), AUC(0-t), t1/2, λz, CL/F and Vd/F are calculated for subjects using non-compartment analysis method.

Physical examination, electrocardiogram and clinical laboratory tests are conducted at screening and 168 hours after administration of each dose; vital signs are measured at scheduled time; adverse events are recorded throughout the study. Clinically relevant safety measurement values are tabulated to evaluate the safety and tolerability of lamotrigine dispersible/chewable tablet. Safety evaluation lasts up to 168 hours after the second oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male non-smoker, based on medical history and physical examination.
* 18-40 years old, inclusive.
* Body weight >50 kg, and result of BMI is between 18.0 and 24.0 kg/m2, inclusive.
* Capable of returning to study site for follow-up according to the requirement of protocol and willing to comply with the policy, procedure and restriction of the study.
* Capable of reading and understanding the information listed in the consent form. Signing the informed consent prior to any study related procedure.
* Results of laboratory tests within the range of reference normal range, or slight abnormality which judged as not clinically significant by investigator.
* AST, ALT, alkaline phosphatase and total bilirubin =<1.5 x ULN ((total bilirubin >1.5 x ULN alone is acceptable if direct bilirubin <35% of total bilirubin).
* Normal blood pressure (systolic blood pressure 90-140 mmHg, diastolic blood pressure < 90mmHg) and pulse rate (60-100/min).
* No clinically significant abnormality on 12-lead ECG.
* Corrected QT interval < 450 ms; or corrected QT interval < 480 ms for subjects with bundle-branch block.
* Male subjects with female partners of child-bearing potential must agree to use contraceptive method after first dose of study treatment and until two weeks after the completion of the study.

Exclusion Criteria:

* Current or chronic history of cardiovascular, respiratory, gastrointestinal, endocrine, hepatic, hematological, psychical or nervous system diseases, use of drug that can change the absorption, metabolism or elimination of study drug, or result in danger or other drugs or diseases that interfere with the interpretation of study data.
* Personal or familial history of hypersensitivity to lamotrigine or drug with similar chemical composition.
* Participation in other clinical trial within 30 days prior to enrollment in the study.
* Use of prescription or non-prescription drugs, including monoamine oxidase inhibitor or herbal drug within 14 days prior to the screening; excluding use of lubricating oil or contraceptive barrier device containing spermicidal agents, and other contraception device.
* History of abnormality of liver function, abnormal hepatic or biliary system, or positive hepatitis B surface antigen (HBsAg), or positive hepatitis C surface antibody (HCAb) or ALT ≥ 2x upper limit of normal (ULN). Having Gilbert syndrome.
* Positive serum HIV antibody.
* Alcohol abuser, defined as alcohol consumption exceeding 3 units/day or 21 units/week. A unit equal to about 240 ml beer, 25 ml spirits or 125 ml wine.
* Positive drug monitoring at screening.
* Evidence for obviously active disease of hematological system, or obvious blood loss within 3 months.
* Blood donation 3 months prior to study.
* Current or past history of nervous-psychiatric disorder, as assessed by Columbia Suicide Severity Rating Scale-baseline evaluation or in the opinion of investigator that the subject is at risk of suicide or with history of suicide behavior/attempt.
* Unsuitable for participating in the study according to the law.
* Unsuitable for participating in the study in the opinion the investigator.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04-28 (Actual); Primary Completion 2013-06-06 (Actual); Study Completion 2013-06-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity [AUC(0-inf)], including bioequivalence evaluation | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  AUC(0-inf) is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-inf) is defined as area under the concentration vs. time curve from zero to infinity.
Area under the concentration-time curve up to the last time point at which the concentration is above the lower limit of quantification [AUC(0-t)], including bioequivalence evaluation | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  AUC(0-t) is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-t) is defined as AUC from time 0 to the last data point above the Lower Limit of Quantification.
The observed maximum serum drug concentration (Cmax), including bioequivalence evaluation | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
Elimination half-time (t½) | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
Elimination rate constant, linear regression according to linear serum drug concentration-time curve | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115207 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115207?search=study&search_terms=115207#rs
- Available data/document: Study Protocol: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register